CLINICAL TRIAL: NCT06700252
Title: Effects of Vestibular Rehabilitation in the Treatment of Dizziness and Balance Disturbances After Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Marschner (Other)
Collaborators: Minot State University (Other)
Responsible Party: Sponsor-Investigator, Beth Marschner, Assistant Professor, Minot State University
Organization: Minot State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2133
Record Dates: First submitted 2024-09-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Concussion
Keywords: Vestibular Rehabilitation; Concussion; Dizziness; Balance Disturbances
MeSH Terms: conditions — Brain Concussion; Dizziness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vestibular Rehabilitation (Experimental): This arm of the study received the vestibular rehabilitation treatment in addition to following traditional protocol.
  Interventions: Other: Vestibular Rehabilitation
- Traditional Treatment (Active Comparator): This arm of the study received the traditional protocol in a stepwise progression only.
  Interventions: Other: Traditional Protocol

INTERVENTIONS:
Other: Vestibular Rehabilitation — This intervention used gaze stabilization, habituation, balance training and exertional training. Exercises utilized included visual tracking, gaze holding with head turns, saccades, visual accommodation exercises, visual convergence exercises, positional accommodation, rockerboard proprioception, single leg balance on the floor and on dynamic surfaces, tandem balance on the floor and on dynamic surfaces, double leg balance on dynamic surfaces, mirror feedback of functional activities, and physical exertion training with walking, biking or sport specific activities.
  Arms: Vestibular Rehabilitation
Other: Traditional Protocol — This intervention symptom management and graduated return to physical activity involving a stepwise progression in which the participant proceeded to the next step if symptom-free at the current step for a 24-hour period. If any symptoms occurred at that step, the participant was returned to the previous step and tried to progress again after 24 hours of rest. The steps were as follows: 1) Patient to return to regular activities such as school 2) Light aerobic activity to increase the patient's heart rate achieved with 5 to 10 minutes on a stationary bike or walking but without weightlifting 3) Moderate activity which increased the heart rate with head or body movement that may have included sport specific exercise with minimal-moderate resistance 4) Heavy, non-contact activity in three planes of movement 5) Full contact practice 6) Competition
  Arms: Traditional Treatment

SUMMARY:
The goal of this clinical trial is to study the effects of including vestibular rehabilitation in the treatment of dizziness and balance disturbances in athletes after concussion. The main questions it aims to answer are:

* Does inclusion of vestibular rehabilitation treatment have an effect on symptom resolution in those with concussion?
* Does inclusion of vestibular rehabilitation treatment have an effect on the rate of recovery and return to play after concussion? Researchers will compare vestibular rehabilitation treatment inclusion in concussion treatment to a traditional concussion treatment approach to see if the rate of symptom resolution and return to play are affected by including vestibular rehabilitation for participants who have experienced a concussion within one week of presenting for the study.

Participants will:

* Be randomly assigned to either receive vestibular rehabilitation included in their concussion treatment or have traditional concussion treatment without vestibular rehabilitation.
* Complete treatment sessions two times per week for up to four weeks
* Complete the corresponding home program for the treatment group
* Complete baseline symptom testing and repeat the symptom testing at study completion for data comparison. Testing includes: Sport Concussion Assessment Tool (SCAT5) including 1) the athlete's background 2) symptom evaluation 3) cognitive screening 4) neurological screening and 5) delayed recall, a Dynamic Gait Index (DGI) including 1) gait on level surface 2) change in gait speed 3) gait with horizontal head turns 4) gait with vertical head turns 5) gait and pivot turn 6) step over obstacle 7) step around obstacle 8) stairs, and a vestibular evaluation including 1) patient history 2) visual assessment 3) vertebral artery clearance 4) cervical spine clearance 5) inner ear assessment 6) brief balance assessment.

DETAILED DESCRIPTION:
Nothing further to include that is not entered or uploaded elsewhere in the record

ELIGIBILITY:
Inclusion Criteria:

* Athlete from a small regional university
* Experiences a concussion
* Identified by their certified athletic trainer to have dizziness or balance dysfunctions
* Referred for initial contact testing and treatment

Exclusion Criteria:

* Acute spinal cord injury with neurological deficits
* Epidural and subdural hematoma with known manifestations
* Acute cervical spine injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Dynamic Gait Index | Up to 4 weeks
  The Dynamic Gait Index (DGI) includes 1) gait on level surface 2) change in gait speed 3) gait with horizontal head turns 4) gait with vertical head turns 5) gait and pivot turn 6) step over obstacle 7) step around obstacle 8) stairs. Each item is scored on a four-point ordinal scale, ranging from 0-3. "0" indicates the lowest level of function, severe impairment and "3" indicates the highest level of function, normal. There are a total of 24 possible points. The lower the score out of 24, the more balance difficulties.
Sport Concussion Assessment Tool 5 | Up to 4 weeks
  The Sport Concussion Assessment Tool 5 includes: athlete's background, symptom evaluation, cognitive screening, neurological screening, and delayed recall. The symptom scale is from 0 (none) to 6 (severe). There are 22 symptoms with a max score of 132. The higher the score, the more severe. The cognitive screening includes 5 orientation questions, immediate memory using recall of 5 word lists, concentration tasks of backward digit recall starting with three digits and progressing to more if able, recalling the months of the year in reverse and delayed recall at the end of the assessment for the immediate memory word list again. The neurological screening assesses reflexes, pupil response and motor function. Balance is examined using the modified balance error scoring system where more errors indicates more balance issues.
Oculomotor Assessment | Up to 4 weeks
  Oculomotor Assessment is used to evaluate eye movement and function to determine if movement and function are normal or abnormal. This includes: smooth pursuits, horizontal saccades, vertical saccades, convergence, vestibulo-ocular reflex (VOR), and visual motion sensitivity Test (VMS).
Semicircular Canal Assessment | Up to 4 weeks
  Semicircular Canal Assessment is used to evaluate how well the inner ear's semicircular canals detect head movement. Tests included in this were the Hallpike-Dix for assessing the posterior canal and the Roll Test for assessing the horizontal canal.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Marschner, DPT, Principal Investigator — Minot State University
Locations (1):
- Minot State University, Minot, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No
The individual participant data is not the main focus of the study. The overall findings of the study with the larger number of participants to look at the trend is what will be shared (presented or published). The IRB proposal for this study included confidentiality of each individual participant as that will be maintained, but the global findings are what will be shared after data analysis for comparison.